CLINICAL TRIAL: NCT05197140
Title: Role of the Protein Matrix in the Anabolic Response to a Ground Beef Patty as Opposed to the Impossible (Vegi-) Burger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 273554
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2023-03

CONDITIONS: Protein Metabolism

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator will be blinded to group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 ounce beef patty (Active Comparator): Subjects consume one beef patty of 4 ounces of cooked meat.
  Interventions: Other: food: cooked 85% lean ground beef
- 4 ounce vegetarian burger (Experimental): Subjects consume one patty of 4 ounces of cooked vegetarian product.
  Interventions: Other: food: Impossible Burger (R)
- 2x 4 ounce vegetarian burger (Experimental): Subjects consume two patties of 4 ounces of cooked vegetarian product.
  Interventions: Other: food: Impossible Burger (R)

INTERVENTIONS:
Other: food: cooked 85% lean ground beef — see arm description
  Other Names: hamburger
  Arms: 4 ounce beef patty
Other: food: Impossible Burger (R) — see arm description
  Other Names: Impossible Burger (R)
  Arms: 2x 4 ounce vegetarian burger; 4 ounce vegetarian burger

SUMMARY:
Several of the investigator's recent studies have shown that all dietary proteins are not equal when it comes to making proteins in human bodies. Generally, foods made from animal muscle tissue are much more efficient at making new proteins in the body that those from plant sources. This study will measure the amount of protein growth in participants after consuming either one beef patty, one vegi-burger, or two vegi-burgers. By using stable isotope infusions and collecting blood and leg muscle samples, the investigator's lab can determine the rate of muscle metabolism that happens after a participant eats a protein-containing food. The investigator wants to determine if the vegi-burger is as efficient as the beef patty at creating proteins in a participants. The investigator will measure this metabolism over a 10-hour period, with the food being eaten at the 4 hour mark. The investigator plans to perform this procedure on up to 8 participants per food option (24 total).

DETAILED DESCRIPTION:
According to the USDA Economic Research Service Food Availability Data, beef consumption has been on a general decline for the past 40 years, with current per capita consumption approximately 35% lower in 2020 than in 1980. Some of this decline over the past few years can be attributed to politically motivated claims that carbon emissions from cattle represent a major threat to the global environment. However, the major reason for declining beef consumption is the widely promulgated claim that beef is unhealthy. The hamburger in particular has become a poster child for the notion that beef consumption is responsible for the increasing occurrence of obesity in the United States. The trend of decreasing beef consumption due to perceived health concerns, particularly obesity and associated health problems, has led major fast-food chains such as Burger King and McDonalds, to offer vegetarian burgers as healthy alternatives to the traditional beef burger. However, examination of the components of the macronutrient matrix of a typical vegetarian burger gives reason to question the health benefits as compared to a traditional beef patty-hamburger.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 40 yrs.
* Body Mass Index of 20-32 inclusive

Exclusion Criteria:

* Unwilling to eat animal proteins
* History of diabetes that requires medication for control of blood glucose
* History of malignancy or chemo/radiation therapy in the 6 months prior to enrollment
* History of gastrointestinal bypass/reduction surgery (Lapband, gastric sleeve, etc.)
* Pregnant females
* Hemoglobin less than 12 g/dL at screening
* Platelets less than 150,000 at screening
* Subjects who cannot refrain from using protein or amino acid supplements for 7 days prior to Visit 3
* Concomitant use of oral or injectable corticosteroids
* Concomitant use of testosterone, IGF-1, or similar anabolic agent
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAMS Center on Aging, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Church DD, Hirsch KR, Kviatkovsky SA, Matthews JJ, Ferrando AA, Azhar G, Wolfe RR. The anabolic response to a ground beef patty and soy-based meat alternative: a randomized controlled trial. Am J Clin Nutr. 2024 Nov;120(5):1085-1092. doi: 10.1016/j.ajcnut.2024.08.030. Epub 2024 Aug 31. PMID 39222687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 Ounce Beef Patty | 4 Ounce Vegetarian Burger | 2x 4 Ounce Vegetarian Burger
Started | 11 | 11 | 11
Completed | 8 | 8 | 8
Not Completed | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 Ounce Beef Patty | 4 Ounce Vegetarian Burger | 2x 4 Ounce Vegetarian Burger | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (7.4) | 36.5 (4.2) | 28.9 (5.8) | 32.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 4 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 7 | 8 | 7 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Plasma Essential Amino Acid Concentration Incremental Area-under-the-curve [ Time Frame: 360 Minutes]
Description: Free leucine, isoleucine, valine, histidine, lysine, methionine, phenylalanine, threonine, tryptophan (combined) (µmol·L^(-1)·min). Following time points (in minutes) post-ingestion will be used to calculate the incremental area under the curve: 60, 90, 120, 180, 210, 240, 270, 300, 330, 360.
Time Frame: 6 hours after consumption of intervention
Measure: Mean (Standard Deviation); unit: micromoles per liter per minute
Arm/Group | 4 Ounce Beef Patty | 4 Ounce Vegetarian Burger | 2x 4 Ounce Vegetarian Burger
Number analyzed (Participants) | 8 | 8 | 8
micromoles per liter per minute | 117896 (45787) | 75098 (45231) | 94058 (27252)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of the study: total 6 months.
Description: Definitions did not differ.
Arm/Group | 4 Ounce Beef Patty | 4 Ounce Vegetarian Burger | 2x 4 Ounce Vegetarian Burger
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT05197140/Prot_SAP_000.pdf